CLINICAL TRIAL: NCT05130190
Title: RAFA Trial: Radiofrequency Ablation of Adenomyosis
Brief Title: Radiofrequency Ablation of Adenomyosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Principal Investigator, Katherine Smith, Assistant Professor of Obstetrics & Gynecology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU-2021-0741
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Adenomyosis
Keywords: adenomyosis; radiofrequency ablation
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RF Treatment (Other): At the time of the subject's trans-abdominal or laparoscopic hysterectomy, the ProVu System will be used to apply RF treatment to one or two adenomas, focal areas of adenomyosis, or diffuse adenomyosis.
  Interventions: Device: RF Treatment

INTERVENTIONS:
Device: RF Treatment — ProVu treatment probe will be energized and RF energy delivered in a pre-programmed, controlled method based on the predetermined size of the affected tissue.
  Other Names: ProVu System

SUMMARY:
To observe the effects of radiofrequency ablation on adenomyosis through the pathological analysis of treated tissue that has been removed during planned hysterectomy.

DETAILED DESCRIPTION:
The ProVu™ System (Hologic, Inc., Boston, MA) is designed and cleared by the FDA as a treatment method for soft tissue, including the treatment of symptomatic uterine fibroids. After locating the general region of the target tissue, a laparoscopic ultrasound transducer is placed on the serosal surface of the uterus to identify the size, location, and number of focal adenomyosis (or adenomyomas). Under ultrasound guidance, the treatment probe (handpiece) is inserted through the serosal surface and into the target tissue. The electrode array containing multiple thermocouples is then deployed according to the size of the target tissue and the position is verified using the ultrasound transducer. Once correctly placed, the surgeon initiates ablation by pressing the foot pedal. Continuous temperature feedback is displayed on the generator screen. For safety purposes, dispersive pads are placed on the patient's thighs to disperse electrical current. If the target tissue is irregular or large, the needle array is retracted and the probe repositioned within the same area under ultrasound guidance. The ablation is repeated until the area of interest is ablated. Overlapping ablations may be required. At the conclusion of the final ablation, the surgeon retracts the array withdraws the probe through the serosal surface of the uterus while coagulating the track to avoid bleeding. Once hemostasis is confirmed and all target tissue has been treated, the surgeon proceeds with the planned hysterectomy and the tissue is examined by a pathologist to assess the ablation zones within the adenomyoma or focal adenomyosis.

ELIGIBILITY:
Inclusion Criteria:

* planning to undergo an abdominal, laparoscopic, or robotic-assisted hysterectomy due to benign conditions
* uterus < 16 weeks gestational size if undergoing a laparoscopic or robotic procedure (no size limit for patients planning to undergo a transabdominal hysterectomy)
* at least one area of focal or diffuse adenomyosis or adenomyomas that is/are contralateral to any fibroids as determined by MRI
* able to provide informed consent
* suitable candidates for surgery (have passed a standard pre-operative health assessment)
* English speaking

Exclusion Criteria:

* require emergent hysterectomy or vaginal hysterectomy
* have a uterus > 16 weeks gestational size if undergoing a laparoscopic or robotic procedure (no size limit for patients planning to undergo a transabdominal hysterectomy)
* have fibroids in the proximity of the target adenomyosis (same side, similar location)
* are not appropriate surgical candidates as determined during pre-operative health assessment
* are unable or unwilling to undergo a hysterectomy
* are pregnant or lactating
* are under the age of 18 years
* have active pelvic inflammatory disease
* have a history of gynecologic malignancy within the past 3 years
* are unable to give informed consent
* have an implantable uterine or fallopian tube device for contraception
* are not English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Post-operative evidence of adenomyoma tissue ablation as assessed by pathological analysis | Day of intervention within 4 hours of RF (radiofrequency) treatment and 2 hours of completion of hysterectomy
  Evidence of ablation to be determined through TTC (Triphenyltetrazolium Chloride) staining with presence of a pink-maroon color change indicating functional enzyme activity and absence of color change indicating non-functional enzyme activity

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kho, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No